CLINICAL TRIAL: NCT01899118
Title: A Multicenter Phase II Trial of Nimotuzumab in Combination With Chemoradiation in Patients With Locally Advanced Rectal Cancer
Brief Title: Nimotuzumab in Combination With Chemoradiation in Patients With Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH-ARO2013
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: locally advanced rectal cancer; Neoadjuvant chemoradiotherapy; Nimotuzumab
MeSH Terms: interventions — nimotuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab plus chemoradiotherapy (Experimental)
  Interventions: Radiation: Preoperative irradiation; Drug: Nimotuzumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Radiation: Preoperative irradiation — 50.4Gy/28F/5.5w
Drug: Nimotuzumab — 400mg/w，0-5w
Drug: Oxaliplatin — 130mg/m2 d1
Drug: Capecitabine — 825mg/m2 bid d1-5/w,1-5w

SUMMARY:
Neoadjuvant (preoperative) concomitant chemoradiotherapy (CRT) is now considered as a standard treatment of locally advanced rectal adenocarcinomas, which correlates better local control and higher sphincter preservation rate. Nimotuzumab, a humanized monoclonal antibody against epidermal growth factor receptor (EGFR) has been reported to improve the therapeutic effect of radiotherapy in some cancers. This study is a clinical phase II trial designed to evaluate the efficacy of the combination of Nimotuzumab administered concurrently with neoadjuvant chemoradiotherapy in patients with locally advanced rectal cancer, and to further investigate its side-effect and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age:18-75 years
3. Histologically confirmed locally advanced colorectal cancer (adenocarcinoma)
4. The lower edge of the tumors located below 12 cm from the anal verge
5. Karnofsky Performance Scale ≥70 points, Life expectancy ≥ 6 months
6. No prior chemotherapy was used
7. No history of regional radiation treatment inthe pelvic cavity
8. Adequate hematologic function: Hb ≥ 100 g/L , WBC≥3.5×109, ANC ≥ 1.5×109 /L，PLT ≥ 100×109 /L Adequate renal function: Cr ≤ 1.5×ULN, TB≤2.5 × ULN Adequate hepatic function: ALT/AST ≤ 2.5×ULN, Alkaline phosphatase ≤ 2.5×ULN
9. Patients without peripheral neuropathy

Exclusion Criteria:

1. Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ
2. Rectal cancer patients with concurrent colon cancer
3. Pregnant or lactating women
4. Fertile female patients without using any contraceptives
5. Allergic to cisplatin and fluorouracil
6. Patients with previous peripheral neuropathy
7. Serious complications: myocardial infarction, heart failure (NYHA Classification>II grade),psychiatric history and severe diabetes
8. Treatment with other anti-cancer therapy(including Chinese herbal medicine)
9. Organ transplant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Pathology complete remission rate | 1 year
  Pathology complete remission rate is the primary outcome measure.

SECONDARY OUTCOMES:
tumor regression rate | 1 year
local recurrence rate | 5 years
overall survival | 5 years
sphincter preservation rate | 3 years
Incidence of Adverse Events | up to 1 month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China